CLINICAL TRIAL: NCT06561035
Title: Opiate Sparing Pain Management Protocol After Anterior Cruciate Ligament Reconstruction Surgery
Brief Title: ACL-R Opioid Sparing Study
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Campbell Clinic (Other)
Responsible Party: Principal Investigator, Joseph Lamplot, Associate Professor, Department of Orthopaedic Surgery and Biomechanical Engineering, Campbell Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-09976-FB
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opiate Sparing (Experimental): Discharge medications:
  1. Medrol Dosepak, take per package instructions from postoperative day 1 to postoperative day 6.
  2. Diclofenac 75 milligram (mg) twice per day from postoperative day 7 to postoperative day 14.
  3. Tylenol 1000 mg three times per day from postoperative day 1 to postoperative day 14.
  4. Gabapentin 100 mg three times per day from postoperative day 1 to postoperative day 14.
  5. Methocarbamol (Robaxin) 750mg twice per day from postoperative day 1 to postoperative day 14.
  6. Promethazine 25 mg every 8 hours as needed for nausea.
  7. Aspirin 81 once per day from postoperative day 1 to postoperative day 30.
  8. Senokot-S (Sennosides and Docusate) as needed for constipation.
  9. 10 tablets of Tramadol 50mg as needed for moderate breakthrough pain only.
  10. 5 tablets of oxycodone 5mg as needed for severe breakthrough pain only.
  11. Supervised physical therapy to start within postoperative day 2 and postoperative day 7.
  Interventions: Drug: Opiate Sparing
- Opiate Based (Active Comparator): Discharge medications:
  1. Diclofenac 75 milligram (mg) twice per day from postoperative day 1 to postoperative day 14.
  2. Tylenol 1000 mg three times per day from postoperative day 1 to postoperative day 14.
  3. Gabapentin 100 mg three times per day from postoperative day 1 to postoperative day 14.
  4. Methocarbamol (Robaxin) 750mg twice per day from postoperative day 1 to postoperative day 14.
  5. Promethazine 25 mg every 8 hours as needed for nausea.
  6. Aspirin 81 once per day from postoperative day 1 to postoperative day 30.
  7. Senokot-S (Sennosides and Docusate) as needed for constipation.
  8. 10 tablets of Tramadol 50mg as needed for moderate breakthrough pain only.
  9. 5 tablets of oxycodone 5mg as needed for severe breakthrough pain only.
  10. Supervised physical therapy to start within postoperative day 2 and postoperative day 7.
  Interventions: Drug: Opiate Based

INTERVENTIONS:
Drug: Opiate Sparing — Subjects will receive medications in the Opiate Sparing arm for pain control.
  Arms: Opiate Sparing
Drug: Opiate Based — Subjects will receive medications in the Opiate Based arm for pain control.
  Arms: Opiate Based

SUMMARY:
This is a randomized control trial to investigate the effectiveness of a multimodal opiate sparing analgesic regimen in controlling post-operative pain and potentially reduce post-operative opioid consumption in patients undergoing Anterior Cruciate Ligament Reconstruction (ACL-R).

DETAILED DESCRIPTION:
There is increased attention on opioid prescription patterns and post-operative narcotic consumption in light of the ongoing opioid crisis in the United States. Patients with opioid use disorders often have their first exposure to opioids following a medical or surgical procedure (Shah et al., 2019). Approximately 6% of patients who were opioid native preoperatively and received opioids postoperatively became long term users. As orthopedic surgeons account for approximately 8% of all dispensed opioid prescriptions (Volkow et al., 2011), surgeons have investigated the effectiveness of multimodal analgesic regimens in controlling post-operative pain and reducing the amount of opioid consumption. Recent studies have shown that an opiate sparing regimen consisted of nonsteroidal anti-inflammatory drugs can control post-operative pain adequately while reducing opioid consumption in patients who underwent arthroscopic knee or shoulder surgeries (Gazendam et al., 2022; Jones et al., 2022). Currently, there is no clear consensus on pain management regimen after anterior cruciate ligament reconstruction.

The purpose of this study is to 1) investigate the difference in pain score and opioid consumption among patients who receive the opioid-based protocol and those who receive opioid-sparing protocol; 2) minimize and potentially eliminate the utilization of narcotics following anterior cruciate ligament reconstruction (ACL-R) surgery.

ELIGIBILITY:
Inclusion Criteria:

* 14-85 years of age.
* Patients undergoing primary ACL-R with or without meniscus repair or meniscectomy, with or without chondroplasty.
* Patients weigh at least 90lbs at time of enrollment.
* Surgery scheduled at a Campbell Clinic Surgery Center (Midtown or Wolf River).
* Willing and able to provide written informed consent.
* Willing and able to cooperate with postoperative therapy.
* Speak and read fluent English.

Exclusion Criteria:

* Multiligament knee reconstruction.
* Pre-injury opioid consumption.
* Substance abuse disorder (illicit drug abuse, alcoholism, etc).
* Concomitant injuries or surgeries warranting pain medication (i.e. polytrauma patient).
* Chronic pain syndrome.
* Renal disease.
* Currently taking selective serotonin reuptake inhibitors and/or serotonin and norepinephrine reuptake inhibitors.
* Known sensitivity, allergy, or intolerance to medications within protocols.
* History of diabetes.
* Currently taking glucagon-like peptide 1 agonist.
* Female patient who is pregnant on day of surgery or becomes pregnant during study period.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Once per day from postoperative day 1 to postoperative day 14; at two weeks follow up visit, 6 weeks follow up visit and 12 weeks follow up visit.
  Record pain score with 0 being no pain at all and 10 being worst pain possible.
Oral morphine equivalent | daily pill count from postoperative day 1 to postoperative day 14; at 2-week follow up visit, 6-week follow up visit and 12-week follow up visit.
  Opiate pill count

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse event. | From day of surgery to 12-week follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lamplot, MD, Principal Investigator — Campbell Clinic
Locations (1):
- Campbell Clinic, Memphis, Tennessee, United States